CLINICAL TRIAL: NCT01802021
Title: Efficacy Study of Chinese Medicine on Modulating Immune Alterations in Advanced Stage, Non-small Cell Lung Cancer Patients Receiving 1st Line Doublet Chemotherapy and 2nd Line Target Therapy
Brief Title: Effect of Astragalus-based Formula: Qingshu-Yiqi-Tang on Modulating Immune Alterations in Lung Cancer Patients
Acronym: QSYQT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 97-1967A3
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2009-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: chinese medicine; non-small cell lung cancer; immunosuppression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qingshu-Yiqi-Tang+standard therapy (Experimental): Plus astragalus-based formula: Qingshu-Yiqi-Tang 7.2gm BID during 1st line chemotherapy and 2nd line target therapy, maximal for 6 months.
  1st line doublet chemotherapy: Cisplatin 70 mg/m2+Taxotere 60 mg/m2 D1/Q3W x 6 cycles, and then 2nd line target therapy: Erlotinib 150mg QD.
  Interventions: Drug: Astagalus-based Formula: Qingshu-Yiqi-Tang
- 1st line doublet chemotherapy (No Intervention): 1st line doublet chemotherapy: Cisplatin 70 mg/m2+Taxotere 60 mg/m2 D1/Q3W x 6 cycles, and then 2nd line target therapy: Erlotinib 150mg QD.

INTERVENTIONS:
Drug: Astagalus-based Formula: Qingshu-Yiqi-Tang — Plus astragalus-based formula: Qingshu-Yiqi-Tang 7.2gm BID during 1st line chemotherapy and 2nd line target therapy.
  maximal for 6 months
  Other Names: Chuang Song Zong Pharmaceutical Co., Ltd. Taiwan.; CHING SHUU YIH CHIH TANG /QING SHU YI QI TANG
  Arms: Qingshu-Yiqi-Tang+standard therapy

SUMMARY:
The myeloid-derived suppressor cells (MDSCs) can further trigger cytotoxic T cell apoptosis, and may shift the macrophages toward M2 subtype, inhibit the Th1 cell, and initiate other immune suppressive mechanism. The functions of NK cells and regulatory T cells are altered, resulting in a disturbance of anti-tumor immune function. All these can further create an environment with a benefit for malignant cell growth and advancement. Astragalus-based formula may confer its survival advantage in cancer patients through modulating the immune system and reversing the immunosuppressive microenvironment.

The investigators aim to study the role of Qingshu-Yiqi-Tang in reversing the immune alterations in patients with advanced stage, non-small cell lung cancer who receive 1st line doublet chemotherapy of cisplatin plus doxetaxel（or Pemetrexed for adenocarcinoma）and 2nd line target therapy of erlotinib. The investigators can explore the possible mechanism of the Astragalus-based formula: Qingshu-Yiqi-Tang in modulating and reversing immunosuppression in advanced stage, non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of mortality and morbidity in the world. In Taiwan, lung cancer is the second cause of cancer death in men and the first in women. Although the five-year survival rate in the early stage, operable non-small cell lung cancer patients was ranged from 60% in stage IA patients to 15% in stage IIIA patients, over 85% of patients were of advanced and inoperable stage at diagnosis. Their medium survival was around six to nine months. New generations of chemotherapy or newly developed target therapy can significantly prolong the medium survival in statistics but the range is only one to three months, which is of limited significance in clinical practice, suggesting a limitation of current modalities of treatment. Chinese herbal medicines have a long history and show effectiveness in benefiting the maintenance of health and the recovery from diseases. Among them, Astragalus-based Chinese herbs have shown to increase effectiveness of platinum-based chemotherapy when combined with chemotherapy in advanced stage non-small cell lung cancer. Despite the fact that many Chinese herbal medicines have shown a pro-apoptotic effect on tumor cells in vitro, none of them have been demonstrated a tumorocidal effect in clinical practice, when used alone. Moreover, Astragalus has revealed an anti-apoptotic effect on cells, suggesting a non-tumorocidal function of Astragalus formula in benefiting cancer therapy.

Studies have shown that external or internal stimuli can induce cell transformation. As a result, dys-regulation in cell growth, DNA repair, cell proliferation and apotosis may occur. Normal committed tissue cells can transform into undifferentiated, multi-potential malignant cells. Normally, the competent immune system can recognize the transformed abnormal cells, undergo immune editing, activate cytotoxic cells to eradicate the abnormal cells and, finally, prevent malignant cell transformation. But through unknown mechanisms, the malignant cells may escape from immune surveillance, release chemokines, growth factors and other mediators to drive the change of inflammatory cells. Consequently, the anti-tumor function of immune cells is suppressed, leading to an environment in favor of development and metastasis of malignant cells. From the experiment of animal model and some observations on malignancy, researchers have suggested that malignant cells can release mediators, which can activate pre-myeloid suppressors and promote myeloid-derived suppressor cells development. The myeloid-derived suppressor cells can further trigger cytotoxic T cell apoptosis, and may shift the macrophages toward M2 subtype, inhibit the Th1 cell, and initiate other immune suppressive mechanism. The functions of NK cells and regulatory T cells are altered, resulting in a disturbance of anti-tumor immune function. All these can further create an environment with a benefit for malignant cell growth and advancement. Astragalus-based formula may confer its surval advantage in cancer patients through modulating the immune system and reversing the immunosuppressive microenvironment.

The lung cancer study in the Department of Thoracic Medicine has demonstrated that the myeloid-derived suppressor cells, cytotoxic T cells, Treg cells and monocytes play a critically important role in mediating immune alterations in patients with advanced stage, non-small cell lung cancer. In this three-year proposal, we aim to study the role of one Astragalus-based formula : Qingshu Yiqi Tang in reversing the immune alterations in patients with advanced stage, non-small cell lung cancer who receive 1st line doublet chemotherapy of cisplatin plus doxetaxel（or Pemetrexed for adenocarcinoma）and 2nd line target therapy of erlotinib. We will target on the modulating effect of Qingshu-Yiqi-Tang on the expression and function of myeloid-derived suppressor cells, Th1, Th2, cytotoxic T cells, NK cells, and the subtypes of monocytes (M1-like vs M2-like). Flow cytometry will be used to study the cell subtypes. The related cytokines and growth factors in serum or supernatant of culture, including IL4, IL-6, IL13, VEGF, TGFb, GM-CSF, will be analyzed using ELISA and FACS microbeads array. The expression of iNOS and arginase I will be verified using WB, IP and RT-PCR. The molecular mechanism related to the cell function will be studied using ex vivo cell co-culture model. All the patients will be followed up for three years at maximum. We hope that, via this three-year proposal, we can explore the possible mechanism of the Astragalus-based formula : Qingshu-Yiqi-Tang(清暑益氣湯) in modulating and reversing immunosuppression in advanced stage, non-small cell lung cancer patients. Through this study, we would found a basis for further comprehensive research on the mechanism of other Chinese herbal medicines for benefiting lung cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathological diagnosis of primary non-small-cell lung cancer Stage IIIB, IV
2. Age ≧ 18 years
3. Written, informed consent
4. ECOG: 0-1

Exclusion Criteria:

1. Subjects with inflammatory, infectious or immune disorder, such as TB, AIDS, active pneumonia, DM, SLE, rheumatoid disease.
2. Subjects with systemic organ disease, such as CHF, ESRD, hepatitis, liver cirrhosis.
3. Subjects with malignancy other than NSCLC.
4. Subjects receiving anti-inflammatory or immunosuppressor medications, such as steroid (oral, except for chemotherapy premedication, or inhaled), NSAIDs.
5. Patients with no willing to sign the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
Progression-free interval | 3 years

OTHER OUTCOMES:
Quality of Life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tse-Hung Huang, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Center for traditional chinese medicine, Chang Gung Memorial Hospital, Gueishan Township, Taoyuan County, Taiwan